CLINICAL TRIAL: NCT05265858
Title: Clinical Phenotypes in Persons With Hip Osteoarthritis and Prognostic Factors for Outcome After Total Hip Arthroplasty
Acronym: HIPPROCLIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Bijzonder onderzoeksfonds (BOF) (Unknown); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Professor, Hasselt University
Other Study IDs: B3712021000002; CTU2020128 (Registry Identifier: Clinical Trial Unit Ziekenhuis Oost-Limburg)
Record Dates: First submitted 2022-02-09; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Hip Osteoarthritis; Total Hip Arthroplasty
Keywords: Hip Osteoarthritis; Total Hip Arthroplasty; Prognostic factors; Pain; Disability; Psychotraumatic events; Fear-Avoidance; Self-efficacy; Perceived Injustice; Quantitative Sensory Testing; Clinical phenotype; Psychopathology
MeSH Terms: conditions — Osteoarthritis, Hip; Pain | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hip osteoarthritis: Patients with hip osteoarthritis who will undergo total hip arthroplasty
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Direct Anterior Approach (DAA) Total Hip Arthroplasty (THA)

SUMMARY:
This prospective longitudinal cohort study aims (1) to identify clinical phenotypes in persons with hip osteoarthritis and after total hip arthroplasty, and (2) to identify prognostic factors for outcomes after total hip arthroplasty.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the leading causes of pain and disability worldwide, with more than 300 million people currently affected by the disease. The hip joint is clinically one of the most affected locations of OA. Each year, more than 40 million prevalent cases and more than 2 million incident cases of hip OA are reported worldwide. The global prevalence and incidence of hip OA are expected to increase considerably in the upcoming decades, as a result of the aging population and an increasing prevalence of risk factors such as obesity and sedentary lifestyle. Since the population with hip OA is highly heterogeneous, individualized care pathways are needed instead of the current one-size-fits-all approach in clinical management. The identification of distinct subgroups within the population with hip OA might offer a foundation for individualized care pathways with the potential improvement of clinical outcomes. Therefore, the first aim of this longitudinal prospective cohort study is to identify clinical phenotypes in persons with hip osteoarthritis based on a set of contributing biopsychosocial variables, and to compare these phenotypes in terms of pain and disability before and after total hip arthroplasty (THA).

Correspondingly with the increasing prevalence and incidence of hip OA, the mean utilization rate of hip implants per 100.000 inhabitants in Organisation for Economic Co-operation and Development (OECD) countries is expected to increase from 145 in 2010 to 275 in 2050. Annually, more than 30.000 THA's are performed in Belgium. This number is growing considerably, especially in younger, working-age patients. Total hip arthroplasty (THA) is a cost-effective procedure in patients with end-stage hip OA. However, previous studies have reported that 8% of patients are dissatisfied with the outcome, and up to 23% of patients report long-term pain after THA. Furthermore, over 30% of patients report activity limitations and about 25% of patients report participation restrictions after THA. An important step towards understanding and improving outcomes after THA is prognostic factor research. Therefore, the second aim of this clinical study is to identify prognostic factors for outcomes of pain and disability after THA in persons with hip OA.

In this prospective longitudinal cohort study, 200 persons undergoing total hip arthroplasty for hip OA will be followed one-year post-surgery. Participants are recruited at the orthopaedic department of 'Ziekenhuis Oost-Limburg' in Genk and at 'de heuppraktijk' in Herselt. Participants will be assessed on a set of biopsychosocial variables, including pain-related fear-avoidance behavior, perceived injustice, psychopathology, traumatic experiences, social support, and self-efficacy. Furthermore, the somatosensory function will be assessed with thermal quantitative sensory testing (QST) and muscle strength will be assessed with a handheld dynamometer (MicroFet 2). Outcome measures include the Hip Disability and Osteoarthritis Outcome Score (HOOS), the OARSI recommended minimum core set of performance-based outcome measures (PBMs), the Patient-Specific Functional Scale (PSFS), Pain intensity (NPRS), Global Perceived Effect (GPE), and satisfaction (NRS). All these measurements will be performed before surgery, as well as 6 weeks, 3 months, and 12 months after surgery. Pain-related fear-avoidance behavior, perceived injustice, anxiety, depression, and pain will be assessed in the early postoperative phase.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a confirmed clinical or radiographic primary diagnosis of hip osteoarthritis who will undergo total hip arthroplasty (THA)

Exclusion Criteria:

* Rheumatoid arthritis or other rheumatic diseases
* Another pathological condition explaining the symptoms (e.g. avascular necrosis)
* Neurological condition (e.g. Parkinson's disease, stroke...) significantly influencing the symptoms of hip osteoarthritis.
* Revision THA
* History of pathological fractures (e.g. osteoporosis, tumor...)
* Contralateral THA during follow-up period
* Total knee arthroplasty (TKA) during follow-up period
* Another surgery planned during follow-up period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with hip osteoarthritis who will undergo THA
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score (HOOS) | 1 week before THA
  The HOOS is a self-reported questionnaire for evaluating symptoms and disability in patients with hip complaints. The questionnaire has been validated in Dutch and consists of 40 items, divided into five subscales: symptoms (5 items), pain (10 items), functioning in activities of daily living (ADL)(17 items), functioning in sport and recreation (4 items), and quality of life (4 items). Each question is scored on a 5-point Likert scale, in which a higher score reflects fewer complaints. A normalized score from 0 to 100 is calculated for the total scale, and for each subscale individually.
Hip disability and Osteoarthritis Outcome Score (HOOS) | 6 weeks after THA
  The HOOS is a self-reported questionnaire for evaluating symptoms and disability in patients with hip complaints. The questionnaire has been validated in Dutch and consists of 40 items, divided into five subscales: symptoms (5 items), pain (10 items), functioning in activities of daily living (ADL)(17 items), functioning in sport and recreation (4 items), and quality of life (4 items). Each question is scored on a 5-point Likert scale, in which a higher score reflects fewer complaints. A normalized score from 0 to 100 is calculated for the total scale, and for each subscale individually.
Hip disability and Osteoarthritis Outcome Score (HOOS) | 3 months after THA
  The HOOS is a self-reported questionnaire for evaluating symptoms and disability in patients with hip complaints. The questionnaire has been validated in Dutch and consists of 40 items, divided into five subscales: symptoms (5 items), pain (10 items), functioning in activities of daily living (ADL)(17 items), functioning in sport and recreation (4 items), and quality of life (4 items). Each question is scored on a 5-point Likert scale, in which a higher score reflects fewer complaints. A normalized score from 0 to 100 is calculated for the total scale, and for each subscale individually.
Hip disability and Osteoarthritis Outcome Score (HOOS) | 12 months after THA
  The HOOS is a self-reported questionnaire for evaluating symptoms and disability in patients with hip complaints. The questionnaire has been validated in Dutch and consists of 40 items, divided into five subscales: symptoms (5 items), pain (10 items), functioning in activities of daily living (ADL)(17 items), functioning in sport and recreation (4 items), and quality of life (4 items). Each question is scored on a 5-point Likert scale, in which a higher score reflects fewer complaints. A normalized score from 0 to 100 is calculated for the total scale, and for each subscale individually.

SECONDARY OUTCOMES:
Patient Specific Functional Scale (PSFS) | 1 week before THA
  The PSFS measures the functional status of the patient. The patient is asked to name the three most important activities for him that are difficult for him or which he is unable to perform because of his problems. Finally, the patient scores the degree of impairment in the activities on an 11-point NRS scale (0-10), where 0 stands for 'cannot perform the activity' and 10 'can perform the activity just as well as before occurrence of the problem'.
Patient Specific Functional Scale (PSFS) | 6 weeks after THA
  The PSFS measures the functional status of the patient. The patient is asked to name the three most important activities for him that are difficult for him or which he is unable to perform because of his problems. Finally, the patient scores the degree of impairment in the activities on an 11-point NRS scale (0-10), where 0 stands for 'cannot perform the activity' and 10 'can perform the activity just as well as before occurrence of the problem'.
Patient Specific Functional Scale (PSFS) | 3 months after THA
  The PSFS measures the functional status of the patient. The patient is asked to name the three most important activities for him that are difficult for him or which he is unable to perform because of his problems. Finally, the patient scores the degree of impairment in the activities on an 11-point NRS scale (0-10), where 0 stands for 'cannot perform the activity' and 10 'can perform the activity just as well as before occurrence of the problem'.
Patient Specific Functional Scale (PSFS) | 12 months after THA
  The PSFS measures the functional status of the patient. The patient is asked to name the three most important activities for him that are difficult for him or which he is unable to perform because of his problems. Finally, the patient scores the degree of impairment in the activities on an 11-point NRS scale (0-10), where 0 stands for 'cannot perform the activity' and 10 'can perform the activity just as well as before occurrence of the problem'.
36-Item Short Form Health Survey (SF-36) | 1 week before THA
  The SF-36 is used to measure perceived health and health-related quality of life. The questionnaire has 36 items containing eight health-related categories: physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, mental health, energy, general health perception, and social functioning. A high score corresponds to a better state of health.
36-Item Short Form Health Survey (SF-36) | 6 weeks after THA
  The SF-36 is used to measure perceived health and health-related quality of life. The questionnaire has 36 items containing eight health-related categories: physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, mental health, energy, general health perception, and social functioning. A high score corresponds to a better state of health.
36-Item Short Form Health Survey (SF-36) | 3 months after THA
  The SF-36 is used to measure perceived health and health-related quality of life. The questionnaire has 36 items containing eight health-related categories: physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, mental health, energy, general health perception, and social functioning. A high score corresponds to a better state of health.
36-Item Short Form Health Survey (SF-36) | 12 months after THA
  The SF-36 is used to measure perceived health and health-related quality of life. The questionnaire has 36 items containing eight health-related categories: physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, mental health, energy, general health perception, and social functioning. A high score corresponds to a better state of health.
Global Perceived Effect (GPE) | 1 day after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 3 days after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 5 days after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 7 days after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 6 weeks after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 3 months after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Global Perceived Effect (GPE) | 12 months after THA
  The patient's opinion about recovery after THA will be measured using the Global Perceived Effect (GPE) score on a 7-point Likert scale, where 1 stands for "a lot worse" and 7 for "a lot better".
Numerical Rating Scale (NRS) of Patient Satisfaction | 1 day after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 3 days after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 5 days after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 7 days after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 6 weeks after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 3 months after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Rating Scale (NRS) of Patient Satisfaction | 12 months after THA
  Patient satisfaction will be measured on an 11-point Numerical Rating Scale (NRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 1 week before THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 1 day after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 3 days after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 5 days after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 7 days after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 6 weeks after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 3 months after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
Numerical Pain Rating Scale (NPRS) | 12 months after THA
  Average pain intensity last week and pain intensity at the moment will be measured on an 11-point Numerical Pain Rating Scale (NPRS), where 0 stands for "no pain" and 10 for "worst imaginable pain".
30-second Chair Stand Test | 1 week before THA
  The 30-second Chair Stand Test will be used to assess sit-to-stand activity (physical function). The maximum number of chair stand repetitions within 30 seconds will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
30-second Chair Stand Test | 6 weeks after THA
  The 30-second Chair Stand Test will be used to assess sit-to-stand activity (physical function). The maximum number of chair stand repetitions within 30 seconds will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
30-second Chair Stand Test | 3 months after THA
  The 30-second Chair Stand Test will be used to assess sit-to-stand activity (physical function). The maximum number of chair stand repetitions within 30 seconds will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
30-second Chair Stand Test | 12 months after THA
  The 30-second Chair Stand Test will be used to assess sit-to-stand activity (physical function). The maximum number of chair stand repetitions within 30 seconds will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
11-step Stair Climb Test | 1 week before THA
  The 11-step Stair Climb Test will be used to assess ascending and descending stair activity (physical function). The time in seconds to ascend and descend 11 stairs will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
11-step Stair Climb Test | 6 weeks after THA
  The 11-step Stair Climb Test will be used to assess ascending and descending stair activity (physical function). The time in seconds to ascend and descend 11 stairs will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
11-step Stair Climb Test | 3 months after THA
  The 11-step Stair Climb Test will be used to assess ascending and descending stair activity (physical function). The time in seconds to ascend and descend 11 stairs will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
11-step Stair Climb Test | 12 months after THA
  The 11-step Stair Climb Test will be used to assess ascending and descending stair activity (physical function). The time in seconds to ascend and descend 11 stairs will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
40-meter (4x10-meter) Fast Paced Walk Test | 1 week before THA
  The 40-meter (4x10-meter) Fast Paced Walk Test will be used to assess short distance walking activity (physical function). The time in seconds to walk 4 x 10 meters for a total of 40 meters will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
40-meter (4x10-meter) Fast Paced Walk Test | 6 weeks after THA
  The 40-meter (4x10-meter) Fast Paced Walk Test will be used to assess short distance walking activity (physical function). The time in seconds to walk 4 x 10 meters for a total of 40 meters will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
40-meter (4x10-meter) Fast Paced Walk Test | 3 months after THA
  The 40-meter (4x10-meter) Fast Paced Walk Test will be used to assess short distance walking activity (physical function). The time in seconds to walk 4 x 10 meters for a total of 40 meters will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).
40-meter (4x10-meter) Fast Paced Walk Test | 12 months after THA
  The 40-meter (4x10-meter) Fast Paced Walk Test will be used to assess short distance walking activity (physical function). The time in seconds to walk 4 x 10 meters for a total of 40 meters will be used as the outcome value. Movement quality during the performance-based tests is assessed based on acceleration data measured with an Inertial Measurement Unit (IMU).

OTHER OUTCOMES:
Thermal Detection and Pain Threshold Temperatures | 1 week before THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the hip) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | 6 weeks after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the hip) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | 3 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the hip) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | 12 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the hip) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Temporal Summation of Pain (TSP) | 1 week before THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | 6 weeks after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | 3 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | 12 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Conditioned Pain Modulation (CPM) | 1 week before THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  * Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  * Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | 6 weeks after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  * Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  * Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | 3 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  * Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  * Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | 12 months after THA
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  * Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  * Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Mini International Neuropsychiatric Interview - Simplified (M.I.N.I.-S for DSM-V) | 1 week before THA
  The MINI-S is a brief structured diagnostic interview for the major psychiatric disorders in the DSM-5. The MINI-S assesses the 17 most common disorders in mental health, including Bipolar Disorder Type 1 and Type 2, Major Depressive Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Generalized Anxiety Disorder, Obsessive Compulsive Disorder, Post-Traumatic Stress Disorder, Acute Stress Disorder, Attention-Deficit/Hyperactivity Disorder, Anorexia Nervosa, Bulimia Nervosa, Alcohol Use Disorder, Substance other than alcohol Use Disorder, Psychotic Disorders.
Mini International Neuropsychiatric Interview - Simplified (M.I.N.I.-S for DSM-V) | 12 months after THA
  The MINI-S is a brief structured diagnostic interview for the major psychiatric disorders in the DSM-5. The MINI-S assesses the 17 most common disorders in mental health, including Bipolar Disorder Type 1 and Type 2, Major Depressive Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Generalized Anxiety Disorder, Obsessive Compulsive Disorder, Post-Traumatic Stress Disorder, Acute Stress Disorder, Attention-Deficit/Hyperactivity Disorder, Anorexia Nervosa, Bulimia Nervosa, Alcohol Use Disorder, Substance other than alcohol Use Disorder, Psychotic Disorders.
Traumatic Experiences Checklist (TEC) | 1 week before THA
  The Traumatic Experiences Checklist (TEC) is a self-reported questionnaire that investigates traumatic experiences in the past. The TEC consists of 31 items, which represent traumatic experiences. Participants should indicate whether they experienced the events and at what age it occurred. The extent to which the event was stressful for the person is also examined. This is scored on a 5-point scale ranging from 'to some extent' to 'to a very severe degree'.
Traumatic Experiences Checklist (TEC) | 12 months after THA
  The Traumatic Experiences Checklist (TEC) is a self-reported questionnaire that investigates traumatic experiences in the past. The TEC consists of 31 items, which represent traumatic experiences. Participants should indicate whether they experienced the events and at what age it occurred. The extent to which the event was stressful for the person is also examined. This is scored on a 5-point scale ranging from 'to some extent' to 'to a very severe degree'.
Childhood Trauma Questionnaire (CTQ) | 1 week before THA
  The CTQ is used to determine whether a person has experienced childhood trauma. The CTQ is a 25-item retrospective self-reported questionnaire that evaluates childhood events. Each question is answered on a 5-point Likert scale (1 never true, 2 often true, 3 sometimes, 4 often true, 5 true). The questionnaire assesses five dimensions of child abuse: (1) Physical abuse, (2) Emotional abuse, (3) Sexual abuse, (4) Physical neglect and (5) Emotional neglect.
Childhood Trauma Questionnaire (CTQ) | 12 months after THA
  The CTQ is used to determine whether a person has experienced childhood trauma. The CTQ is a 25-item retrospective self-reported questionnaire that evaluates childhood events. Each question is answered on a 5-point Likert scale (1 never true, 2 often true, 3 sometimes, 4 often true, 5 true). The questionnaire assesses five dimensions of child abuse: (1) Physical abuse, (2) Emotional abuse, (3) Sexual abuse, (4) Physical neglect and (5) Emotional neglect.
Hospital Anxiety and Depression Scale (HADS) | 1 week before THA
  The HADS is a 14-item questionnaire evaluating anxiety and depression complaints without involving physical complaints. The HADS consists of two subscales, one subscale covers symptoms of anxiety (HADS-A), the other symptoms of depression (HADS-D). Each item is scored from zero ("not applicable") to three ("certainly applicable"). The maximum score on each subscale is 21, with higher values indicating more anxiety/depression symptoms.
Hospital Anxiety and Depression Scale (HADS) | 1 week after THA
  The HADS is a 14-item questionnaire evaluating anxiety and depression complaints without involving physical complaints. The HADS consists of two subscales, one subscale covers symptoms of anxiety (HADS-A), the other symptoms of depression (HADS-D). Each item is scored from zero ("not applicable") to three ("certainly applicable"). The maximum score on each subscale is 21, with higher values indicating more anxiety/depression symptoms.
Hospital Anxiety and Depression Scale (HADS) | 6 weeks after THA
  The HADS is a 14-item questionnaire evaluating anxiety and depression complaints without involving physical complaints. The HADS consists of two subscales, one subscale covers symptoms of anxiety (HADS-A), the other symptoms of depression (HADS-D). Each item is scored from zero ("not applicable") to three ("certainly applicable"). The maximum score on each subscale is 21, with higher values indicating more anxiety/depression symptoms.
Hospital Anxiety and Depression Scale (HADS) | 3 months after THA
  The HADS is a 14-item questionnaire evaluating anxiety and depression complaints without involving physical complaints. The HADS consists of two subscales, one subscale covers symptoms of anxiety (HADS-A), the other symptoms of depression (HADS-D). Each item is scored from zero ("not applicable") to three ("certainly applicable"). The maximum score on each subscale is 21, with higher values indicating more anxiety/depression symptoms.
Hospital Anxiety and Depression Scale (HADS) | 12 months after THA
  The HADS is a 14-item questionnaire evaluating anxiety and depression complaints without involving physical complaints. The HADS consists of two subscales, one subscale covers symptoms of anxiety (HADS-A), the other symptoms of depression (HADS-D). Each item is scored from zero ("not applicable") to three ("certainly applicable"). The maximum score on each subscale is 21, with higher values indicating more anxiety/depression symptoms.
Fear-Avoidance Component Scale (FACS) | 1 week before THA
  Pain-related fear avoidance was assessed by the Dutch version of the FACS, which is a 20-item questionnaire, with each item scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five fear-avoidance-related severity levels have been proposed: subclinical (0 to 20), mild (21 to 40), moderate (41 to 60), severe (61 to 80), and extreme (81 to 100).
Fear-Avoidance Component Scale (FACS) | 1 week after THA
  Pain-related fear avoidance was assessed by the Dutch version of the FACS, which is a 20-item questionnaire, with each item scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five fear-avoidance-related severity levels have been proposed: subclinical (0 to 20), mild (21 to 40), moderate (41 to 60), severe (61 to 80), and extreme (81 to 100).
Fear-Avoidance Component Scale (FACS) | 6 weeks after THA
  Pain-related fear avoidance was assessed by the Dutch version of the FACS, which is a 20-item questionnaire, with each item scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five fear-avoidance-related severity levels have been proposed: subclinical (0 to 20), mild (21 to 40), moderate (41 to 60), severe (61 to 80), and extreme (81 to 100).
Fear-Avoidance Component Scale (FACS) | 3 months after THA
  Pain-related fear avoidance was assessed by the Dutch version of the FACS, which is a 20-item questionnaire, with each item scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five fear-avoidance-related severity levels have been proposed: subclinical (0 to 20), mild (21 to 40), moderate (41 to 60), severe (61 to 80), and extreme (81 to 100).
Fear-Avoidance Component Scale (FACS) | 12 months after THA
  Pain-related fear avoidance was assessed by the Dutch version of the FACS, which is a 20-item questionnaire, with each item scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five fear-avoidance-related severity levels have been proposed: subclinical (0 to 20), mild (21 to 40), moderate (41 to 60), severe (61 to 80), and extreme (81 to 100).
Tampa Scale for Kinesiophobia (TSK-17) | 1 week before THA
  Pain-related fear of movement was assessed with the 17-item version of the TSK. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement.
Tampa Scale for Kinesiophobia (TSK-17) | 1 week after THA
  Pain-related fear of movement was assessed with the 17-item version of the TSK. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement.
Tampa Scale for Kinesiophobia (TSK-17) | 6 weeks after THA
  Pain-related fear of movement was assessed with the 17-item version of the TSK. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement.
Tampa Scale for Kinesiophobia (TSK-17) | 3 months after THA
  Pain-related fear of movement was assessed with the 17-item version of the TSK. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement.
Tampa Scale for Kinesiophobia (TSK-17) | 12 months after THA
  Pain-related fear of movement was assessed with the 17-item version of the TSK. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement.
Injustice Experience Questionnaire (IEQ) | 1 week before THA
  Perceived injustice was measured with the Injustice Experience Questionnaire (IEQ). The IEQ consists of 12 items, each item is scored from zero ("not at all") to four (all the time"). The total score ranges between 0 and 48 and higher total scores reflect higher levels of perceived injustice.
Injustice Experience Questionnaire (IEQ) | 1 week after THA
  Perceived injustice was measured with the Injustice Experience Questionnaire (IEQ). The IEQ consists of 12 items, each item is scored from zero ("not at all") to four (all the time"). The total score ranges between 0 and 48 and higher total scores reflect higher levels of perceived injustice.
Injustice Experience Questionnaire (IEQ) | 6 weeks after THA
  Perceived injustice was measured with the Injustice Experience Questionnaire (IEQ). The IEQ consists of 12 items, each item is scored from zero ("not at all") to four (all the time"). The total score ranges between 0 and 48 and higher total scores reflect higher levels of perceived injustice.
Injustice Experience Questionnaire (IEQ) | 3 months after THA
  Perceived injustice was measured with the Injustice Experience Questionnaire (IEQ). The IEQ consists of 12 items, each item is scored from zero ("not at all") to four (all the time"). The total score ranges between 0 and 48 and higher total scores reflect higher levels of perceived injustice.
Injustice Experience Questionnaire (IEQ) | 12 months after THA
  Perceived injustice was measured with the Injustice Experience Questionnaire (IEQ). The IEQ consists of 12 items, each item is scored from zero ("not at all") to four (all the time"). The total score ranges between 0 and 48 and higher total scores reflect higher levels of perceived injustice.
General Self-Efficacy Scale (GSES) | 1 week before THA
  The General Self-Efficacy Scale is a self-reported questionnaire used to measure self-efficacy. The GSES measures how a person generally copes with stressors/difficult situations in life. It consists of ten statements (optimistic "self-beliefs") that ask about how people think and act in general. Items are scored on a 4-point Likert scale.
General Self-Efficacy Scale (GSES) | 6 weeks after THA
  The General Self-Efficacy Scale is a self-reported questionnaire used to measure self-efficacy. The GSES measures how a person generally copes with stressors/difficult situations in life. It consists of ten statements (optimistic "self-beliefs") that ask about how people think and act in general. Items are scored on a 4-point Likert scale.
General Self-Efficacy Scale (GSES) | 3 months after THA
  The General Self-Efficacy Scale is a self-reported questionnaire used to measure self-efficacy. The GSES measures how a person generally copes with stressors/difficult situations in life. It consists of ten statements (optimistic "self-beliefs") that ask about how people think and act in general. Items are scored on a 4-point Likert scale.
General Self-Efficacy Scale (GSES) | 12 months after THA
  The General Self-Efficacy Scale is a self-reported questionnaire used to measure self-efficacy. The GSES measures how a person generally copes with stressors/difficult situations in life. It consists of ten statements (optimistic "self-beliefs") that ask about how people think and act in general. Items are scored on a 4-point Likert scale.
Groningen Orthopaedic Social Support Scale (GO-SSS) | 1 week before THA
  The 'Groningen Orthopedic Social Support Scale' is a self-reported questionnaire that has been developed to measure social support in patients with a THA or TKP. Social support is measured through 12 statements where the patient can choose from four answers: 'never or rarely', 'occasionally', 'regularly' or 'often'.
Groningen Orthopaedic Social Support Scale (GO-SSS) | 6 weeks after THA
  The 'Groningen Orthopedic Social Support Scale' is a self-reported questionnaire that has been developed to measure social support in patients with a THA or TKP. Social support is measured through 12 statements where the patient can choose from four answers: 'never or rarely', 'occasionally', 'regularly' or 'often'.
Groningen Orthopaedic Social Support Scale (GO-SSS) | 3 months after THA
  The 'Groningen Orthopedic Social Support Scale' is a self-reported questionnaire that has been developed to measure social support in patients with a THA or TKP. Social support is measured through 12 statements where the patient can choose from four answers: 'never or rarely', 'occasionally', 'regularly' or 'often'.
Groningen Orthopaedic Social Support Scale (GO-SSS) | 12 months after THA
  The 'Groningen Orthopedic Social Support Scale' is a self-reported questionnaire that has been developed to measure social support in patients with a THA or TKP. Social support is measured through 12 statements where the patient can choose from four answers: 'never or rarely', 'occasionally', 'regularly' or 'often'.
Muscle strength | 1 week before THA
  Hip muscle strength will be measured with the MicroFet 2®, a handheld dynamometer. In the test protocol, each muscle group will be tested three times, with the best value of the three tests as the final result. The following muscle groups will be tested:
  * Hip flexors
  * Hip abductors
  * Hip extensors
  * Hip external rotators
  * Hip adductors
Muscle strength | 6 weeks after THA
  Hip muscle strength will be measured with the MicroFet 2®, a handheld dynamometer. In the test protocol, each muscle group will be tested three times, with the best value of the three tests as the final result. The following muscle groups will be tested:
  * Hip flexors
  * Hip abductors
  * Hip extensors
  * Hip external rotators
  * Hip adductors
Muscle strength | 3 months after THA
  Hip muscle strength will be measured with the MicroFet 2®, a handheld dynamometer. In the test protocol, each muscle group will be tested three times, with the best value of the three tests as the final result. The following muscle groups will be tested:
  * Hip flexors
  * Hip abductors
  * Hip extensors
  * Hip external rotators
  * Hip adductors
Muscle strength | 12 months after THA
  Hip muscle strength will be measured with the MicroFet 2®, a handheld dynamometer. In the test protocol, each muscle group will be tested three times, with the best value of the three tests as the final result. The following muscle groups will be tested:
  * Hip flexors
  * Hip abductors
  * Hip extensors
  * Hip external rotators
  * Hip adductors
Perceived stress | 1 week before THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 1 day after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 3 days after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 5 days after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 7 days after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 6 weeks after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 3 months after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.
Perceived stress | 12 months after THA
  Perceived stress will be evaluated with a single question of the Perceived Stress Scale (PSS): 'During the past day, how often have you felt nervous and stressed?'. The question is scored on a 5-point Likert scale, from 0 'never' to 4 'very often'.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, Principal Investigator — Hasselt University; Kristoff Corten, Principal Investigator — Ziekenhuis Oost-Limburg; Katleen Bogaerts, Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Heuppraktijk, Herselt, Antwerpen
  - Ziekenhuis Oost-Limburg, Genk, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sergooris A, Verbrugghe J, Bonnechere B, Matheve T, Corten K, Bogaerts K, Timmermans A. Inter-individual differences in early post-operative pain, cognitions, and emotions after total hip arthroplasty: A longitudinal cohort study. Clin Rehabil. 2025 Jun;39(6):784-795. doi: 10.1177/02692155251333537. Epub 2025 Apr 21. PMID 40255065
- [Derived] Sergooris A, Verbrugghe J, Matheve T, Van Den Houte M, Bonnechere B, Corten K, Bogaerts K, Timmermans A. Clinical phenotypes and prognostic factors in persons with hip osteoarthritis undergoing total hip arthroplasty: protocol for a longitudinal prospective cohort study (HIPPROCLIPS). BMC Musculoskelet Disord. 2023 Mar 25;24(1):224. doi: 10.1186/s12891-023-06326-9. PMID 36964541